CLINICAL TRIAL: NCT04191213
Title: Efficacy of Gum Arabic as Anti-oxidant, Anti-inflammatory and Fetal Hemoglobin Inducing Agent in Sickle Cell Anemia Patients : A Randomized, Double-blind, Two-armed Parallel-group, Placebo-controlled Phase II/III Study - Khartoum, Sudan
Brief Title: Gum Arabic as Anti-oxidant, Anti-inflammatory and Fetal Hemoglobin Inducing Agent in Sickle Cell Anemia Patients
Acronym: GA&SCA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Neelain University (Other)
Collaborators: University of Khartoum (Other)
Responsible Party: Principal Investigator, Lamis Kaddam, Director, Al-Neelain University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GA& Sickle among children
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Sickle Cell Anemia in Children
Keywords: sickle cell anemia; Gum Arabic; Fetal Hemoglobin
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia | interventions — Gum Arabic; Pectins

STUDY DESIGN:
Intervention Model Description: The intervention group will receive Gum Arabic. And The placebo group will receive pectin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, Investigator and outcome assessor will be masked regarding the type of intervention each group will receive
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This arm will receive 100% natural Gum Arabic provided in a powder form in 30-grams-dose for participants above 5 years of age and 15-grams-dose for participants below 5 years of age for 12 weeks
  Interventions: Dietary Supplement: Acacia Senegal extract
- Control group (Placebo Comparator): This group will be provided with pectin powder provided as one-gram-dose for children below 5 years of age & two-gram-dose for children above 5 years of age
  Interventions: Dietary Supplement: Pectin

INTERVENTIONS:
Dietary Supplement: Acacia Senegal extract — Oral Digestion of Gum Arabic to be consumed early morning in daily basis for 12 weeks
  Other Names: (Gum Arabic)
  Arms: Intervention Group
Dietary Supplement: Pectin — Oral Digestion of Pectin to be consumed early morning in daily basis for 12 weeks
  Arms: Control group

SUMMARY:
To study the efficacy of Gum Arabic as an anti-oxidant, anti-inflammatory and Fetal Hemoglobin-inducing agent among Sickle Cell Disease children. Half of participants will receive Gum Arabic and the other half will receive placebo

DETAILED DESCRIPTION:
Polymerized hemoglobin is injurious to the red cell membrane, resulting in oxidative damage in sickle cell disease . Fetal hemoglobin is protective against sickling and its decrease is associated with vaso-occlusive crisis . Gum Arabic is soluble fibers with prebiotic properties. It increased the level of serum butyrate which is short chain fatty acid. The latter proved to serve as fetal hemoglobin inducing agent both in vivo and in vitro study. And also has strong anti-inflammatory properties. So our aim to test whether oral digestion of Gum Arabic will induce fetal hemoglobin among sickle cell pediatric patients

ELIGIBILITY:
Inclusion Criteria:

* Homozygous for Sickle Cell Disease (SS) as documented by Haemoglobin electrophoresis.

Subjects whom medications and dosages had been stable for 2 weeks before study entry.

Subjects who have not received blood transfusion or had acute episode related to sickle cell disease in the last two weeks before the start of intervention.

Exclusion Criteria:

* Patients with history of Gum Arabic allergy. Patients who have ischemic heart disease, liver dysfunction or hepatitis. Pregnant female patients who plan to conceive in the next 4 months and fertile female patients who are not using an effective contraception method.

Patients who are currently using Gum Arabic. Patients who are on steroids or chemotherapy.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Fetal hemoglobin level after 12 weeks | 12 weeks
  Measure increase from the baseline values
Total anti oxidant capacity | 12 weeks
  Measure increase from the baseline values

SECONDARY OUTCOMES:
Anti inflammatory marker C reactive Protein | 12 weeks
  Measure decrease from the baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Imad M Fdl-Elmula, PhD, Study Director — Alneelain University
Locations (1):
- Military Hospital, Omdurman, Khartoum State, Sudan

IPD SHARING:
Plan to Share IPD: Undecided
Share patients data without personal data and without breaching confidentiality

REFERENCES:
- [Background] Kaddam L, FdleAlmula I, Eisawi OA, Abdelrazig HA, Elnimeiri M, Lang F, Saeed AM. Gum Arabic as fetal hemoglobin inducing agent in sickle cell anemia; in vivo study. BMC Hematol. 2015 Dec 29;15:19. doi: 10.1186/s12878-015-0040-6. eCollection 2015. PMID 26719803
- [Background] Kaddam L, Fadl-Elmula I, Eisawi OA, Abdelrazig HA, Salih MA, Lang F, Saeed AM. Gum Arabic as novel anti-oxidant agent in sickle cell anemia, phase II trial. BMC Hematol. 2017 Mar 16;17:4. doi: 10.1186/s12878-017-0075-y. eCollection 2017. PMID 28331623
- [Background] Kamal E, Kaddam LA, Dahawi M, Osman M, Salih MA, Alagib A, Saeed A. Gum Arabic Fibers Decreased Inflammatory Markers and Disease Severity Score among Rheumatoid Arthritis Patients, Phase II Trial. Int J Rheumatol. 2018 Jul 5;2018:4197537. doi: 10.1155/2018/4197537. eCollection 2018. PMID 30112005